CLINICAL TRIAL: NCT04669379
Title: Preoperative Optimization of Patient's Expectations by the Use of an Online-Tool - a Randomized Controlled Trial
Brief Title: Is an Online-tool Capable of Improving Patients' Outcomes After Surgery?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor, Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Online-Tool Erwartungen prä-OP
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Patients Undergoing Surgery
Keywords: Expectations; Preoperative intervention; placebo effect; surgery; clinical trial; recovery; online intervention

STUDY DESIGN:
Intervention Model Description: The patients will be randomly distributed to the intervention group (IG/EXPECT) or the control group (CG). The intervention group will receive a psychological preoperative online-intervention to optimize expectations. The control group will receive no intervention at all.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG/EXPECT) (Experimental)
  Interventions: Behavioral: EXPECT: Preoperative optimization of patient's expectations
- Standard of Care (SOC) (No Intervention)

INTERVENTIONS:
Behavioral: EXPECT: Preoperative optimization of patient's expectations — Patients work through an online-tool (around 30 minutes). This preoperative intervention aims to optimize patients' expectations by focusing on positive and realistic expectations regarding the surgery-benefits and recovery process, giving information, and giving advice for coping resources.
  Arms: Intervention group (IG/EXPECT)

SUMMARY:
Recovery after the surgery depends on psychological factors such as preoperative information, expectations, and surgery-associated anxiety. Prior studies have shown that even short preoperative psychological interventions can improve postoperative outcomes. However, the content of these interventions needs further examination. This study aims to examine if the developed preoperative intervention (i) reduces preoperative anxiety, (ii) increases positive expectations, and (iii) improves the long-term outcome and postoperative recovery. Therefore an online-tool has been developed. Using an online-approach makes it possible to reach many patients taking as little time and cost as possible.

Patients who undergo surgery in the next two weeks and want to participate in the study will be asked for the planned surgical procedure. There will be a filter (stratum) for surgery. Patients with the same kind of surgery are randomized into two groups (Control vs. intervention group) after they've filled some questionnaires at the baseline assessment. Following this, the intervention group will participate in the psychological online intervention (around 30 minutes). The intervention will focus on the treatment outcome expectations and personal control expectations to increase patients' positive expectations. The control group will receive no psychological intervention. Both groups will fill out questionnaires again in the evening, two days before the surgery, around one week after the surgery, and three months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* In-patient operation under general anesthetic
* Age 18 or above
* Fluency in German
* Informed consent

Exclusion Criteria:

* Participation in other research programs: in agreement with Coordinating Investigator patient can participate substudies, if this do not interfere with the main study
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Change in Pain Disability Index (PDI) from Baseline to two days pre-surgery to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 0 (no disability at all) - 10 (total disability). Consequently higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in The Amsterdam Preoperative Anxiety and Information Scale (APAIS) from Baseline to two days pre-surgery | Baseline, two days pre-surgery
  Items range from 1 (not at all) - 5 (extremely). Higher scores mean patients are more interested in information and do have greater worries
Change in Health Related Quality of Life (Short Form 12, SF-12) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  There are different item scales. The item scale of the first item (General health perceptions) ranges from 1 (excellent)to 5 (bad). The item scales of the second and third item (limitations in physical activities because of health problems)range from 1 (yes, absolutely restricted) to 2 (yes, a bit restricted) to 3 (no, not restricted at all). The item scales of the items 4-7 (limitations in usual role activities because of physical health or emotional problems) are just "yes" and"no". The item scale of the eighth item (bodily pain) ranges from 1 (Absolutely not) to 5 (a lot). The item scales of the items 9-12 (general mental health, vitality and limitations in social activities because of physical or emotional problems)range from 1 (always) to 5 (never).
Change in Patient health questionnaire screener (PHQ) from Baseline to one week post-surgery to three months post-surgery | Baseline, two days pre-surgery, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (not at all) - 4 (nearly everyday). Consequently higher scores mean a worse outcome.
Change in The Primary Appraisal Secondary Appraisal questionnaire (PASA) from Baseline to two days pre-surgery to one week post-surgery | Baseline, two days pre-surgery, up to one week post-surgery, up to three months post-surgery
  Items range from 0 (absolutely wrong) - 6 (absolutely right). Higher scores mean a better outcome.
Change in The Control Attitudes Scale-Revised (CAS-R) from Baseline to one week post-surgery | Baseline, up to one week post-surgery
  Items range from 0 (not at all) - 8 (absolutely right). Higher scores mean a better outcome (after reversion of the inverse items 5 and 8).

OTHER OUTCOMES:
Change in Patients' Illness Perception (Brief Illness Perception Questionnaire, B-IPQ) from Baseline to two days pre-surgery to one week post-surgery to three months after surgery | Baseline, two days pre-surgery, up to one week post-surgery, up to three months post-surgery
  The B-IPQ surveys the cognitive and emotional representations of illness. Item 1-5 measure cognitive illness representations (consequences, timeline, personal control, treatment control, and identity). Item 6 and 8 quantify emotional representations (concern & emotions). Item 7 assesses illness comprehensibility. Item 9 is an open question(three most important causal factors in their illness). Items range from 0-10: item 1: no disability at all to very strong disability, item 2: really short to forever, item 3: no control at all zo extreme control, item 4: not at all to extremely helpful, item 5: no complaints at all to very much and strong complaints, item 6: no worries at all to extreme worries,item 7: not at all to very clear, item 8: emotionally not included at all to emotional extremely included.
Change in patients' expectations (Expected Illness Perception Questionnaire, IPQ-E) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (absolutely wrong) - 5 (absolutely right). Higher scores mean a better outcome.
Change in patients optimism (Life-Orientation-Test Revised, LOT-R) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (absolutely) - 5 (absolutely not). Higher scores mean a worse outcome.
Personality (Big Five Inventory, BFI-10) | Baseline
  Items range from 1 (disagree strongly) - 5 (agree strongly). The questionnaire includes the scales "openness to experience", "conscientiousness", "extraversion", agreeableness and neuroticism
Patients' experience with prior surgeries | Baseline
  Rating of experience with own prior surgeries. Rating of experience with surgeries of close others. First patients are asked if they or close others had a prior surgery before (yes/no). If they answer yes, they are asked to rate their or their close others experience (item ranges from 1 (very bad) - 5 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Clinical Psychology and Psychotherapy Dept. of Psychology, Philipps-University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Auer CJ, Glombiewski JA, Doering BK, Winkler A, Laferton JA, Broadbent E, Rief W. Patients' Expectations Predict Surgery Outcomes: A Meta-Analysis. Int J Behav Med. 2016 Feb;23(1):49-62. doi: 10.1007/s12529-015-9500-4. PMID 26223485
- [Background] Gaab, J. (2009). PASA - Primary Appraisal Secondary Appraisal - Ein Fragebogen zur Erfassung von situationsbezogenen kognitiven Bewertungen, Verhaltenstherapie,19:114-115
- [Background] Juergens MC, Seekatz B, Moosdorf RG, Petrie KJ, Rief W. Illness beliefs before cardiac surgery predict disability, quality of life, and depression 3 months later. J Psychosom Res. 2010 Jun;68(6):553-60. doi: 10.1016/j.jpsychores.2009.10.004. Epub 2009 Dec 5. PMID 20488272
- [Background] Laferton JA, Kube T, Salzmann S, Auer CJ, Shedden-Mora MC. Patients' Expectations Regarding Medical Treatment: A Critical Review of Concepts and Their Assessment. Front Psychol. 2017 Feb 21;8:233. doi: 10.3389/fpsyg.2017.00233. eCollection 2017. PMID 28270786
- [Background] Löwe, B., Spitzer, R. L., Zipfel, S., & Herzog, W. (2002). PHQ-D Gesundheitsfragebogen für Patienten (German Version of the Patient Health Questionnaire). Karlsruhe: Pfizer.
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Moser DK, Riegel B, McKinley S, Doering LV, Meischke H, Heo S, Lennie TA, Dracup K. The Control Attitudes Scale-Revised: psychometric evaluation in three groups of patients with cardiac illness. Nurs Res. 2009 Jan-Feb;58(1):42-51. doi: 10.1097/NNR.0b013e3181900ca0. PMID 19092554
- [Background] Rief, W., & Glombiewski, J. A. (2016). Erwartungsfokussierte Psychotherapeutische Interventionen (EFPI). Verhaltenstherapie, 26(1), 47-54.
- [Background] Rief W, Shedden-Mora MC, Laferton JA, Auer C, Petrie KJ, Salzmann S, Schedlowski M, Moosdorf R. Preoperative optimization of patient expectations improves long-term outcome in heart surgery patients: results of the randomized controlled PSY-HEART trial. BMC Med. 2017 Jan 10;15(1):4. doi: 10.1186/s12916-016-0767-3. PMID 28069021
- [Background] Salzmann, S., Laferton, J., Auer, C., Shedden-Mora, M., Wambach, K., & Rief, W. (2018). Patientenerwartungen optimieren: Beschreibung einer präoperativen Kurzintervention am Beispiel von Patienten vor einer Bypass-Operation. Verhaltenstherapie, 28(3), 157-165.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Rammstedt, B. und O. P. John, 2007: Measuring personality in one minute orless: A 10-item short version of the Big Five Inventory in English and German.Journal of Research in Personality 41: 203-212